CLINICAL TRIAL: NCT04208880
Title: ACAR Brain Health Intervention Study: A Preliminary Investigation of Subjective Memory and Well-Being
Brief Title: ACAR Brain Health Intervention Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Alabama, Tuscaloosa (Other)
Responsible Party: Principal Investigator, Ian M. McDonough, Assistant Professor, University of Alabama, Tuscaloosa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ACARTBH
Record Dates: First submitted 2019-12-18; First posted 2019-12-23 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Aging Well
Keywords: Subjective Memory; Intervention; Brain Health; Educational Program; Well-being

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of six groups in parallel for the duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- TBH Brain Workout 1.0 (Experimental): The TBH Brain Workout program will cover education topics that encourage engagement in interventions shown to impact cognitive performance, including those to enhance intellectual (e.g., how to focus attention), physical (e.g., how to eat healthy), and socio-emotional (e.g., how to stay socially engaged) well-being. The challenge activities will be easy to master.
  Interventions: Behavioral: TBH Brain Workout 1.0
- TBH Brain Workout 2.0 (Experimental): The TBH Brain Workout program will cover education topics that encourage engagement in interventions shown to impact cognitive performance, including those to enhance intellectual (e.g., how to focus attention), physical (e.g., how to eat healthy), and socio-emotional (e.g., how to stay socially engaged) well-being. The challenge activities will be moderately difficult to master.
  Interventions: Behavioral: TBH Brain Workout 2.0
- TBH Memory 1.0 (Experimental): The TBH Memory program will cover educational topics on how memory works, what environmental factors impact memory, and memory strategies. The challenge activities will be easy to master.
  Interventions: Behavioral: TBH Memory 1.0
- TBH Memory 2.0 (Experimental): The TBH Memory program will cover educational topics on how memory works, what environmental factors impact memory, and memory strategies. The challenge activities will be moderately difficult to master.
  Interventions: Behavioral: TBH Memory 2.0
- Book Club (Active Comparator): The Book Club will be given a book to read on how to improve brain health and will discuss separate chapters across 8 sessions. These sessions will be led by the participants and no formal structure will be provided. No personal challenges will be asked of participants and no log will be required. All groups will have a sign-in sheet to record individual participation.
  Interventions: Behavioral: Brain Health Book Club
- No Contact Wait List (No Intervention): The Wait List group will simply take the the surveys at each time point as the other groups.

INTERVENTIONS:
Behavioral: TBH Brain Workout 1.0 — TBH Brain Workout program with easy challenge activities.
  Arms: TBH Brain Workout 1.0
Behavioral: Brain Health Book Club — Each week a new chapter will be read that contains new information to enhance brain health.
  Arms: Book Club
Behavioral: TBH Brain Workout 2.0 — TBH Brain Workout program with moderately difficult challenge activities.
  Arms: TBH Brain Workout 2.0
Behavioral: TBH Memory 1.0 — TBH Memory program with easy challenge activities.
  Arms: TBH Memory 1.0
Behavioral: TBH Memory 2.0 — TBH Memory program with moderately difficult challenge activities
  Arms: TBH Memory 2.0

SUMMARY:
The main objective of this study is to assess the effectiveness of four Total Brain Health educational programs, TBH Brain Workout (1.0 and 2.0) and TBH Memory (1.0 and 2.0), in older adults residing in independent living facilities through the Acts Center for Applied Research (ACAR). Each TBH program trains for lifestyle intervention skills across the wellness spectrum shown by research to promote cognitive performance and reduce dementia risk, using social-based training methods, and experiential learning activities. Each TBH program also has two levels of difficulty (1.0 and 2.0), which will be assessed in independent groups. Each independent living community will administer one TBH program at a time such that participants will be randomly assigned to one of three categories: 1) one of the four educational programs, 2) an active book club that will read and discuss on tips to improve one's brain health, and 3) a wait-list control group. All groups other than the wait-list control group will have 8 sessions across 2 months. The older adults who agree to be a part of the research will be asked to fill out a survey at pre-intervention, post-intervention 1 (immediate), and post-intervention 2 (2 months). We predict that the participants in the TBH Brain Workout and TBH Memory programs (all difficulty levels) will have a greater knowledge about brain health, improved subjective appraisals of their memory, improved social outcomes, lower depression, and reduced dementia risk compared with the two control groups. The investigators predict that the active book club control will differ on brain health knowledge than the wait-list control group. Due to the more cognitively challenging nature of the harder TBH programs, the investigators also predicted that the harder versions would have greater improvement in brain health knowledge and improved subjective appraisals of their memory than the easier versions.

DETAILED DESCRIPTION:
Current evidence suggests that behavioral lifestyle modifications may improve everyday cognitive performance, thereby reducing dementia risk. The main objective of this study is to assess the effectiveness of four Total Brain Health educational programs, TBH Brain Workout (1.0 and 2.0) and TBH Memory (1.0 and 2.0), in older cognitively independent adults residing in independent living facilities through the Acts Center for Applied Research (ACAR). Each TBH program trains skills across the wellness spectrum demonstrated to impact cognitive risk, use social-based training methods, and has experiential learning activities. Each of the two TBH educational programs has two levels of difficulty. The TBH Brain Workout program will consist of 8 sessions that covers topics to encourage engagement in interventions shown to impact cognitive performance, including those to enhance intellectual (e.g., how to focus attention), physical (e.g., how to eat healthy), and socio-emotional (e.g., how to stay socially engaged) well-being. The TBH Memory program will consist of 8 sessions that covers education on how memory works, what environmental factors impact memory, and memory strategies. Participants in both TBH programs will be guided through activities with a trainer, but also will have active learning activities that will include teaching others (collaborative learning), competitive teams, and whole class activities. The more challenging versions of each program (level 2.0) will also include "challenge" activities that encourage them to engage daily in an activity that requires movement, an activity that requires giving thanks, or an activity than requires mental stimulation. Participants will log which challenge activities they engaged in each week. The Book Club will be given a book to read on how to improve brain health and will discuss separate chapters across 8 sessions. These sessions will be led by the participants and no formal structure will be provided. No personal challenges will be asked of participants and no log will be required. All groups will have a sign-in sheet to record individual participation.

Each independent living community will administer one TBH program at a time such that participants will be randomly assigned to one of three categories: 1) one of the four educational programs, 2) an active "book club" that will read and discuss on tips to improve one's brain health, and 3) a wait-list control group. The older adults who agree to be a part of the research will be asked to fill out a survey at pre-intervention, post-intervention 1 (immediate), and post-intervention 2 (2 months). We predict that the participants in the TBH Brain Workout and TBH Memory programs (all difficulty levels) will have a greater knowledge about brain health, improved subjective appraisals of their memory, improved social outcomes, lower depression, and reduced dementia risk compared with the two control groups. We predict that the active book club control will differ on brain health knowledge than the wait-list control group. Due to the more cognitively challenging nature of the harder TBH programs, we also predicted that the harder versions would have greater improvement in brain health knowledge and improved subjective appraisals of their memory than the easier versions.

Power was calculated using the Bias- and Uncertainty-Corrected Sample Size (BUCCS) R package. This package was used because it allowed us to use effect sizes from a pilot study while considering bias and uncertainty in finding a similar effect size. Our pilot study used pre and post-test data from the Brain Health Fund of Knowledge Questionnaire (one of our primary outcome measures) in which we combined two active intervention groups that had earlier versions of the Total Brain Workout 1.0 and Memory 1.0 classes. The pilot data resulted in an F-value of 18.50 (effect size f = .56) from 67 total participants. Our alpha level was set to .0025 to consider a) new recommendations to set a generic alpha level to .005 and b) multiple comparisons corrections for our two primary outcome variables (i.e., Brain Health Fund of Knowledge Questionnaire and Potential for Improvement). The level of assurance and power was set to .8. Using two time points with these parameters, it was estimated that the investigators would need 49 participants per group to detect a significant effect.

Our plan is to recruit at least 49 participants from each of the six groups (four active and two control) through the through ACAR. Participation will be open for all independent living residents from January 2018 to January 2020. Participants will be aged 60 and older who have not been diagnosed with a memory disorder and are not currently engaging in other cognitive or brain training research. If the investigators are unable to reach our recruitment goals by January 2020, they will average together the 1.0 and 2.0 groups within each TBH program to achieve our desired sample size.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 and older

Exclusion Criteria:

* Diagnosed with a memory disorder
* Currently engaging in other cognitive or brain training research

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 294 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Brain Health Fund of Knowledge Questionnaire | 2 months
  Test of knowledge of lifestyle factors that improve brain health, ranging from 0 to 30 with a higher score representing better knowledge.
Memory Controllability Inventory: Potential for Improvement (Lachman, 1995) | 2 months
  Self-reported assessment of one's own potential to improve their own cognition with a minimum score of 3 and maximum of 21 with higher scores indicating greater potential for improvement.

SECONDARY OUTCOMES:
TBH Brain Workout Groups: Center for Epidemiological Survey-Depression (Radloff, 1977) | 2 months
  Self-reported assessment of depressive symptoms, ranging from 0 to 60 where higher scores indicate more depression.
TBH Brain Workout Groups: Daily Habits Questionnaire | 2 months
  Self-reported assessment of engagement in daily activities that promote brain health, ranging from 30 to 210 where higher scores represent more engagement in daily health habits.
TBH Memory Groups: Multifactorial Memory Questionnaire (Troyer & Rich, 2002) | 2 months
  Self-reported assessment of subjective memory on contentment (ranging from 9-72), ability (ranging from 0-77), and strategy (ranging from 9-64) with higher scores being better.
All Groups: Brain Health Fund of Knowledge Questionnaire | 4 months
  Test of knowledge of lifestyle factors that improve brain health, ranging from 0 to 30 with a higher score representing better knowledge.
All Groups: Memory Controllability Inventory: Potential for Improvement (Lachman, 1995) | 4 months
  Self-reported assessment of one's own potential to improve their own cognition with a minimum score of 3 and maximum of 21 with higher scores indicating greater potential for improvement.

OTHER OUTCOMES:
All Groups: Modifiable Dementia Risk Questionnaire (based on Deckers et al., 2015) | 2 and 4 month time points
  Self-report of having modifiable risk factors for dementia, ranging from -5.92 to 13.7 where higher is representative of a greater risk for dementia
All Groups: Revised UCLA Loneliness Scale (Hughes et al., 2004) | 2 and 4 month time points
  Self-report assessment of loneliness, ranging from 17 to 68 where higher numbers represent greater loneliness.
All Groups: The Social Disconnectedness Scale (Cornwell et al., 2009) | 2 and 4 month time points
  Self-report assessment of amount of social support, ranging from 9 to 36 where higher numbers represent greater social support.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Alabama, Tuscaloosa, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cornwell EY, Waite LJ. Social disconnectedness, perceived isolation, and health among older adults. J Health Soc Behav. 2009 Mar;50(1):31-48. doi: 10.1177/002214650905000103. PMID 19413133
- [Background] Deckers K, van Boxtel MP, Schiepers OJ, de Vugt M, Munoz Sanchez JL, Anstey KJ, Brayne C, Dartigues JF, Engedal K, Kivipelto M, Ritchie K, Starr JM, Yaffe K, Irving K, Verhey FR, Kohler S. Target risk factors for dementia prevention: a systematic review and Delphi consensus study on the evidence from observational studies. Int J Geriatr Psychiatry. 2015 Mar;30(3):234-46. doi: 10.1002/gps.4245. Epub 2014 Dec 12. PMID 25504093
- [Background] Hughes ME, Waite LJ, Hawkley LC, Cacioppo JT. A Short Scale for Measuring Loneliness in Large Surveys: Results From Two Population-Based Studies. Res Aging. 2004;26(6):655-672. doi: 10.1177/0164027504268574. PMID 18504506
- [Background] Lachman, M. E., Bandura, M., Weaver, S. L., & Elliott, E. (1995). Assessing memory control beliefs: The memory controllability inventory. Aging, Neuropsychology, and Cognition, 2(1), 67-84.
- [Background] Orgeta V, Mukadam N, Sommerlad A, Livingston G. The Lancet Commission on Dementia Prevention, Intervention, and Care: a call for action. Ir J Psychol Med. 2019 Jun;36(2):85-88. doi: 10.1017/ipm.2018.4. PMID 31187723
- [Background] Radloff, L. S. (1977). The CES-D scale: A self-report depression scale for research in the general population. Applied psychological measurement, 1(3), 385-401.
- [Background] Rosenberg A, Ngandu T, Rusanen M, Antikainen R, Backman L, Havulinna S, Hanninen T, Laatikainen T, Lehtisalo J, Levalahti E, Lindstrom J, Paajanen T, Peltonen M, Soininen H, Stigsdotter-Neely A, Strandberg T, Tuomilehto J, Solomon A, Kivipelto M. Multidomain lifestyle intervention benefits a large elderly population at risk for cognitive decline and dementia regardless of baseline characteristics: The FINGER trial. Alzheimers Dement. 2018 Mar;14(3):263-270. doi: 10.1016/j.jalz.2017.09.006. Epub 2017 Oct 19. PMID 29055814
- [Background] Troyer AK, Rich JB. Psychometric properties of a new metamemory questionnaire for older adults. J Gerontol B Psychol Sci Soc Sci. 2002 Jan;57(1):P19-27. doi: 10.1093/geronb/57.1.p19. PMID 11773220
- [Background] Risk Reduction of Cognitive Decline and Dementia: WHO Guidelines. Geneva: World Health Organization; 2019. Available from http://www.ncbi.nlm.nih.gov/books/NBK542796/ PMID 31219687